CLINICAL TRIAL: NCT03199365
Title: Tu Salud ¡Si Cuenta! Reaching Latino Family Dyads to Increase Physical Activity and Healthy Eating
Brief Title: Tu Salud Si Cuenta Intervention in Increasing Physical Activity and Healthy Eating Among Latino Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-0735; NCI-2018-01136 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0735 (Other: M D Anderson Cancer Center); P30CA016672 (NIH); R56HL128705 (NIH)
Record Dates: First submitted 2017-06-23; First posted 2017-06-26 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (TSSC intervention) (Experimental): Participants undergo two TSSC intervention sessions delivered at participants' homes by trained CHWs over 1.5 hours.
  Interventions: Behavioral: Behavioral Dietary Intervention; Behavioral: Behavioral Intervention

INTERVENTIONS:
Behavioral: Behavioral Dietary Intervention — Undergo TSSC intervention sessions
Behavioral: Behavioral Intervention — Undergo TSSC intervention sessions
  Other Names: Behavior Conditioning Therapy; behavior modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; BEHAVIORAL THERAPY; Behavioral Treatment; Behavioral Treatments

SUMMARY:
This trial studies how a program to encourage healthy behaviors (Tu Salud Si Cuenta) works to increase physical activity and healthy eating habits among Latino families. Improving physical activity and healthy eating habits may help in preventing cancer-related diseases and lead to a better quality of life among Latino families.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conduct formative research with adult Latino family dyads to assess the home environment and current behaviors, and identify perceived determinants of healthy eating and physical activity (PA) within the family context.

II. Adapt the "Tu Salud Si Cuenta" (TSSC) intervention to focus on increasing physical activity (PA) and healthy eating among adult Latino family dyads (TSSC-Family).

III. Evaluate the acceptability of intervention content, materials, and procedures with adult Latino family dyads.

OUTLINE:

FORMATIVE RESEARCH: To adapt the intervention, participants undergo immersive assessment over 3 hours which is conducted by research staff and involves examination of the home food and PA environments, objective and self-reported PA, nutritional intake, demographics and relevant psychosocial measures. Participants are also instructed to wear an accelerometer device to measure physical activity for up to 7 days and participate in in-depth interviews over 1.5 hours.

PRE-TESTING: Participants undergo two TSSC intervention sessions delivered at participants' homes by trained community health workers (CHWs) over 1.5 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported Hispanic/Latino ethnicity
2. Age 18-65 years
3. Speak English or Spanish
4. Physically able to engage in low-to-moderate PA
5. Consumption of fewer than 5 servings of fruits and vegetables per day
6. Valid home address in the Houston neighborhoods of Gulfton, the East End/Magnolia, or Near Northside, or adjacent neighborhoods
7. Working telephone number

Exclusion Criteria:

1) Pregnancy at any point during the study period OR considering pregnancy during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Identification of perceived determinants of healthy eating and physical activity (PA) as determined by questionnaires and interviews | Up to 2 years
  The appropriate summary statistics will be calculated for continuous and categorical variables along with corresponding liberal (i.e., 80%) confidence intervals where appropriate. Boxplots, histograms, and other graphical displays will also be generated in order to describe the sample. Descriptive information will be used to inform future trials aimed at testing the intervention.
Evaluate and adapt the "Tu Salud Si Cuenta" (TSSC/Your Health Matters!) intervention | Up to 2 years
  Results from the formative research phase will inform the adaptation of the TSSC intervention to focus on dyadic collaboration and support. In general, TSSC-Family is proposed as a 6-month intervention involving six monthly home visits by a community health worker (CHW) who will deliver the TSSC curricula (Fitness for Life and Nutritious Eating), adapted for the dyadic approach, using non-directive motivational techniques. Participants will be instructed in standard behavioral skills such as self-monitoring, goal setting, problem solving, and relapse prevention.
Evaluate the acceptability of intervention content, materials, and procedures | Up to 2 years
  The appropriate summary statistics will be calculated for continuous and categorical variables along with corresponding liberal (i.e., 80%) confidence intervals where appropriate. Boxplots, histograms, and other graphical displays will also be generated in order to describe the sample. Descriptive information will be used to inform future trials aimed at testing the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Larkin Strong, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org